CLINICAL TRIAL: NCT06496802
Title: Prognostic Significance of Preoperative Nutritional Status for Postoperative Acute Kidney Injury in Elderly Patients Undergoing Lung Resection Surgery
Brief Title: Prognostic Significance of Preoperative Nutritional Status on Postoperative Acute Kidney Injury
Status: Not yet recruiting | Type: Observational
Sponsor: Wanmin Liao (Other)
Responsible Party: Sponsor-Investigator, Wanmin Liao, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: 101662
Record Dates: First submitted 2024-07-04; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Acute Kidney Injury; Pneumonectomy
Keywords: Acute Kidney Injury; lung resection surgery; malnutrition; prediction model
MeSH Terms: conditions — Acute Kidney Injury; Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
The incidence of postoperative acute kidney injury (AKI) is high in patients undergoing lung resection surgery, especially in the elderly. Early identification of high-risk postoperative AKI patients can help develop prevention and treatment management strategies.

DETAILED DESCRIPTION:
The goal of this retrospective study is to investigate the predictive value of preoperative nutritional status, as measured by three scoring systems - the geriatric nutritional risk index (GNRI), prognostic nutritional index (PNI), and controlling nutritional status (CONUT) score - on postoperative AKI in elderly patients under lung resection surgery.

ELIGIBILITY:
Inclusion Criteria:

1. aged ≥ 65 years
2. lung resection surgery including：pneumonectomy , bilobectomy , lobectomy, segmentectomy, wedge resection/bullectomy.

Exclusion Criteria:

1. patients with an American Society of Anesthesiologists (ASA) physical status V.
2. those with end-stage renal disease (i.e. a glomerular filtration rate of 15 mL/min/1.73 m2 or receiving haemodialysis).
3. those did not have sufficient data required for nutritional evaluation or AKI evaluation.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Older patients (aged ≥ 65 years) who underwent lung resection surgery under general anesthesia at our Hospital between January 2020 and June 2024 were included in our study. Lung resection surgery included pneumonectomy , bilobectomy , lobectomy, segmentectomy, wedge resection/bullectomy.
Sampling Method: Non-Probability Sample
Enrollment: 1880 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2024-09-15 (Estimated); Study Completion 2024-09-15 (Estimated)

PRIMARY OUTCOMES:
Postoperative acute kidney injury | Within 7 days after surgery
  In accordance with the KDIGO creatinine criteria: a serum creatinine increases of 26.5 mmol/L within 48 hours or 1.5 times baseline within 7 days after surgery.

IPD SHARING:
Plan to Share IPD: No